CLINICAL TRIAL: NCT00474110
Title: Ketamine and Hydromorphone PCA Analgesia for Antineoplastic-Induced Pediatric Mucositis
Brief Title: Ketamine and Hydromorphone for Patient Controlled Pain Relief in Children's Mucositis
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Clinical practice had changed between time of initial protocol development and subject recruitment. We were not able to find eligible patients.
Sponsor: University of British Columbia (Other)
Responsible Party: Dr Carolyne Montgomery, University of British Columbia
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H06-03799
Record Dates: First submitted 2007-05-14; First posted 2007-05-16 (Estimated); Last update posted 2010-11-01 (Estimated); Status verified 2010-10

CONDITIONS: Mucositis
Keywords: Ketamine; hydromorphone; pediatric mucositis
MeSH Terms: conditions — Mucositis | interventions — Ketamine; Hydromorphone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Ketamine and hydromorphone for patient-controlled relief in children's mucositis.
  Interventions: Drug: Ketamine & hydromorphone

INTERVENTIONS:
Drug: Ketamine & hydromorphone — See Detailed Description

SUMMARY:
The treatment of cancer in children may result in an extremely painful condition called oral mucositis when the cells lining the mouth are injured due to the cancer medication. Patients with this condition are often unable to take anything by mouth or to swallow their own saliva. This severe pain may last for as long as 2 weeks. A survey of our previous 22 patients showed high daily pain scores despite the use of intravenous (given through a small tube in a vein) opioid medications (family of pain relieving drugs, e.g. morphine and hydromorphone).

The purpose of this pilot study is to determine which of 3 concentrations of ketamine to combine with hydromorphone to provide the best pain relief with minimum side effects. The results from this study will allow us to do a larger study to compare the best concentration found from this study to standard treatment. If successful, this combination of ketamine and hydromorphone will also be used to treat other pain problems in children.

DETAILED DESCRIPTION:
The purpose of this observational pilot study is to evaluate the feasibility, efficacy and optimum ratio of a compounded mixture of HM-K administered parenterally by PCA in pediatric mucositis patients who have inadequate analgesia using conventional HM PCA.

An open-label study of 20 consecutive consenting/assenting subjects who meet the study criteria will be conducted. All patients who are eligible for the study will be approached for informed, written consent and subjects over age 7 will complete an assent form.

The subject will be examined by a pediatric oncology fellow/staff to determine the level of clinical severity of the mucositis using the Oral Mucositis Assessment Scale (OMAS) and World Health Organization Mucositis Scale.

A modified Colour Analogue Scale (mCAS) that was originally designed to evaluate pain intensity will be used to evaluate the self-report symptoms. The subject will then receive 24 hours of therapy using a compounded HM-K PCA solution.

Initial PCA prescription for the Background and Bolus will be set at the existing settings on the morning of recruitment as per the study entry criteria of minimum hourly use of 4 mcg/kg/hour of HM. The 1-hour Maximum will be set at 4 times the Background dose.

At 24 hours, the 24-hour HM and K consumption will be calculated. The subject will be re-examined by a pediatric oncology fellow/staff to determine the level of clinical severity of the mucositis and the self-report symptom evaluation questionnaire administered. Conventional Therapy of HM PCA will be restarted and at 24 hours, both the mucositis severity and the self-report symptom evaluation questionnaire administered. Descriptive summaries of the demographic data will be provided. The 24-hour HM utilization will be compared to the study entry-level utilization (24 hour period prior to recruitment). A 30% reduction in opioid use will be considered clinically important.A Symptom Index of Start Study Symptom Level - End Study Symptom Level / Start Study Symptom level will be calculated for each symptom including pain intensity. An Index of greater than or equal to 0.5 will be considered a positive outcome. Indexes at 0, 24 and 48 hours will be compared. A descriptive summary of the incidence and treatment of opioid-induced side effects at 0, 24 and 48 hours will be provided.

Ketamine Solution Concentrations

Solution 1 (low): HM 0.2 and K 0.2 mg/mL (1:1) - 20 mg/20 mg in 100 mL. Solution 2 (medium): HM 0.2 and K 0.6 mg/mL (1:3) - 20 mg/60 mg in 100 mL. Solution 3 (high): HM 0.2 and K 1 mg/mL (1:5) - 20 mg/100 mg in 100 mL.

The starting solution will be Solution 2 in a minimum dose 4 mcg/kg/hour of hydromorphone (HM) and 12 mcg/kg/hour of ketamine (K) (0.02 mL/kg/hour of solution.

"Add background": 4 mcg/kg/hour of Hydromorphone equivalent (0.02 mL/kg/hour of solution) may occur once as required after solution change criteria are met.

"Increase background": additional 4 mcg/kg/hour of Hydromorphone equivalent (0.02 mL/kg/hour of solution).

Repeat "Increase background": 4 mcg/kg/hour of Hydromorphone equivalent (0.02 mL/kg/hour of solution) may occur 3 hourly as required after solution change criteria are met.

"Decrease background": decrease by 4 mcg/kg/hour of Hydromorphone equivalent (0.02 mL/kg/hour of solution) may occur 3 hourly as required after solution change criteria are met.

"Stop background": Background is stopped so that only bolus dose remains. May occur when background has been reduced to 4 mcg/kg/hour of Hydromorphone for at least 3 hours or exceessive ADEs.

"D/C background: Discontinue background HM and only bolus remains.

"Stop Study (SS)": Converting the PCA to conventional HM therapy with any adjuvants required according to existing practice of Acute Pain Service. For compassionate reasons, if a patient/family expresses a with to remain on STudy Therapy, this will be accepted.

Once patient has ADEs and requires Solution 1, they may not re-start solution 2 or 3.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric oral mucositis due to anti-neoplastic therapy.

Exclusion Criteria:

* Must not be receiving concurrent oral analgesics or sedatives such as acetaminophen, gabapentin, lorazepam, nabilone or clonidine.

Ages: 5 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2009-08; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
24 hour hydromorphone consumption

SECONDARY OUTCOMES:
Self-report symptom scores

CONTACTS AND LOCATIONS:
Overall Officials: Carolyne Montgomery, MD, Principal Investigator — University of British Columbia; Mark Ansermino, MD, Study Director — University of British Columbia; Caron Strahlendorf, MD, Study Director — University of British Columbia; Robert Purdy, MD, Study Director — University of British Columbia; Colleen Court, MD, Study Director — University of British Columbia; Joanne Lim, Study Director — University of British Columbia
Locations (1):
- BC Children's Hospital, Vancouver, British Columbia, Canada